CLINICAL TRIAL: NCT02765789
Title: Immunoadsorption in Anti-glomerular Basement Membrane Glomerulonephritis; a Pilot Study
Brief Title: Immunoadsorption in Anti-GBM Glomerulonephritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, dr. C.F.M. Franssen, Nephrologist, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201500361
Record Dates: First submitted 2016-05-03; First posted 2016-05-09 (Estimated); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Anti-glomerular Basement Membrane Glomerulonephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunoadsorption (Experimental): Immunoadsoprtion (Immunosorba). All (anticipated) 8 participants will be treated with immunoadsorption
  Interventions: Device: Immunoadsorption (Immunosorba)

INTERVENTIONS:
Device: Immunoadsorption (Immunosorba) — Immunoadsorption as an alternative to plasma exchange

SUMMARY:
Anti-glomerular basement membrane (GBM) glomerulonephritis is a rare autoimmune disease mediated by anti-GBM antibodies and characterized by acute renal failure due to diffuse crescentic glomerulonephritis. Established treatment is cyclophosphamide and corticosteroids to suppress anti-GBM production and daily plasma exchange to remove circulating anti-GBM antibodies. The vast majority of patients with anti-GBM glomerulonephritis develop irreversible end-stage renal failure despite this treatment. Immunoadsorption may lower anti-GBM titres more effectively than plasma exchange. The goal of this interventional open, non-randomized pilot study is to study the efficacy, adverse events, logistic feasibility and costs of immuno-adsorption for the removal of anti-GBM antibodies in patients with acute renal failure due to anti-GBM glomerulonephritis. Eight patients with acute renal failure due to anti-GBM glomerulonephritis with or without accompanying pulmonary involvement will be treated with daily immunoadsorption, instead of plasma exchange, until anti-GBM titres are undetectable. All other aspects of the treatment (e.g. immunosuppressive treatment, renal replacement therapy) will be standard. The primary study parameter is the number of days that anti-GBM antibody titre is above a toxic level, defined as >30 ELISA units. Secondary study parameters are the tolerability and adverse events of immunoadsorption, the logistic feasibility defined as the time interval between diagnosis and start of first immunoadsorption treatment and costs of immunoadsorption.

DETAILED DESCRIPTION:
Rationale: Anti-glomerular basement membrane (anti-GBM) glomerulonephritis is a rare organ-specific autoimmune disease that is mediated by anti-GBM antibodies. It is characterized by acute renal failure due to diffuse crescentic glomerulonephritis, often accompanied by pulmonary hemorrhage. Established treatment is cyclophosphamide and corticosteroids to suppress anti-GBM production and daily plasma exchange to remove circulating anti-GBM antibodies. The vast majority of patients with anti-GBM glomerulonephritis develop irreversible end-stage renal failure despite this treatment. The treatment goal in anti-GBM glomerulonephritis is to achieve undetectable anti-GBM titres as rapid as possible. Immunoadsorption is an extracorporeal technique that selectively removes antibodies and may lower anti-GBM titres more effectively than plasma exchange. With this technique the patient's plasma is passed through an immunoadsorption column that contains protein A that binds antibodies of the IgG class like anti-GBM antibodies. However, data on the efficacy of anti-GBM removal by immunoadsorption compared with plasma exchange are scarce. In the literature, there are only a few case descriptions of the clinical effect of immunoadsorption in patients with anti-GBM disease with some cases showing recovery of renal function despite unfavourable prognosis (serum creatinine >500 µmol/l and/or high percentage of crescents on renal biopsy). Immunoadsorption is presently not used in the Netherlands for anti-GBM disease.

Objective: To study the efficacy, adverse events, logistic feasibility and costs of immuno-adsorption for the removal of anti-GBM antibodies in patients with acute renal failure due to anti-GBM glomerulonephritis.

Study design: Interventional, open, non-randomized, pilot study. After informed consent, patients will be treated according to the current treatment protocol with the exception of daily immunoadsorption instead of daily plasma exchange.

Study population: 8 patients with acute renal failure due to anti-GBM glomerulonephritis with or without accompanying pulmonary involvement.

Intervention: Participating patients will be treated with daily immunoadsorption (2.5 times the plasma volume), instead of plasma exchange, until anti-GBM titres are undetectable. All other aspects of the treatment (e.g. immunosuppressive treatment, renal replacement therapy) will be standard.

Main study parameters/endpoints: The primary study parameter is the number of days that anti-GBM antibody titre is above a toxic level, defined as >30 ELISA units. Plasma levels of anti-GBM will be measured before and after each immunoadsorption treatment. Courses of anti-GBM titres will be compared with an historical cohort of patients with anti-GBM disease treated with plasma exchange. Secondary study parameters are: 1. Tolerability and adverse events of immunoadsorption. 2. Logistic feasibility defined as the time interval between diagnosis and start of first immunoadsorption treatment; 3. Costs of immunoadsorption (personnel and materials).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: From a patient's perspective, the burden of daily immunoadsorption is comparable with that of daily plasma exchange with regard to vascular access (central venous catheter) and blood sampling to monitor treatment response. The treatment time is approximately one hour longer than plasma exchange (4 hours instead of 3 hours). Possible adverse effects of immunoadsorption are part of the current study proposal but previous studies in other patient groups suggest that frequency and severity of adverse effects of immunoadsorption are comparable with plasma exchange.

ELIGIBILITY:
Inclusion Criteria:

* Acute renal failure due to anti-GBM glomerulonephritis with or without pulmonary involvement. Eligible patients must have a clinical picture met rapidly progressive glomerulonephritis in combination with one of the following:

  1. Serological evidence of circulating anti-GMB antibodies (Dotblot, Phadia, ELISA). Patients with dual autoantibody positivity (anti-GBM antibodies and ANCA) can participate in this study. 2. Renal biopsy with necrotising glomerulonephritis with linear fluorescence for IgG along the GBM.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Number of days that anti-GBM antibody titre is above a toxic level, defined as >30 ELISA units. | 60 days after study start
  Nr of Days that anti-GBM title is >30 units

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 60 days after study start
  NR of participants with adverse event
Logistic feasibility defined as the time interval between diagnosis and start of first immunoadsorption treatment. | 60 days
  Time interval between diagnosis and start of first immunoadsorption treatment
Costs of immunoadsorption (personnel and materials). | 60 days
  Costs of immunoadsorption treatment

CONTACTS AND LOCATIONS:
Overall Officials: Casper FM Franssen, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Gromiongen, Netherlands

IPD SHARING:
Plan to Share IPD: No